CLINICAL TRIAL: NCT06626893
Title: Integrative "Omics" Approaches for Leukemia Target Identification and Matched Therapeutic Intervention
Acronym: AL-TOMICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Benedetta Cambò, MD, PhD, Azienda Ospedaliero-Universitaria di Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3070
Record Dates: First submitted 2024-03-21; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Myeloid Leukemia, Acute; Leukemia, Acute Lymphoblastic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed Refractory Acute Leukemias (Other): Functional and genomics analyses will be performed on primary sample from each enrolled patient (biological preclinical study)
  Interventions: Biological: Functional tests; Genetic: Next Generation Sequencing analysis; Biological: Microvesicles analysis

INTERVENTIONS:
Biological: Functional tests — Functional analyses will be performed on primary sample from each enrolled patient. Isolated blast cells are cultered and incubated with a specific library of drugs (175 drugs) at four different concentrations for 72 hours.
Genetic: Next Generation Sequencing analysis — For each patient, sequencing analyses will be performed on blast cells (for somatic mutations) and on epithelial cells from buccal swab (for germline mutations)
Biological: Microvesicles analysis — Analyses on microvesicles isolated from both Bone Marrow samples and Peripheral Blood Samples will be performed to investigate the microenvironment of the disease.

SUMMARY:
The goal of this clinical trial is to use multiple "omics" sciences to more thoroughly investigate Acute Recurrent/Refractory Leukemias (LA R/R) after conventional therapy in order to identify new targets and/or therapeutic approaches, in patients with a diagnosis of Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia/ Lymphoblastic Lymphoma B(ALL-B), Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma T (ALL-T), Acute Biphenotypic Leukemia/II as defined by WHO( World Health Organization) 2016, relapsed or refractory after at least one line of therapy. The main question that the trial aims to answer is: "Can molecules with known biological activity be active and represent possible new therapeutic strategies in relapsed/refractory Acute Leukemias on the basis of response profiles identified through the integration of next-generation chemogenomic and functional analyses? " It is expected that a minimum of 100 patients, male and female, aged 18 years and older, will be included. To participate in the study, the patient must consent to the performance on biological specimen (peripheral blood and bone marrow) of genetic/molecular and/or "omics" investigations performed with modern sequencing techniques, such as Next Generation Sequencing, Single Cell RNA Seq (scRNAseq), RT-qPCR(Quantitative reverse transcription polymerase chain reaction). These investigations will aim to improve the understanding of the genetic and molecular alterations of her disease. In addition, your cells will be used in the laboratory to perform in vitro sensitivity studies (drug response profiling - DRP) that aim to simultaneously test a set of hundreds of drugs to assess sensitivity or resistance profiles of your disease cells with the aim of identifying specific new therapies that target specific cellular mechanisms. In addition, part of the biological sample will be used for investigations of the bone marrow microenvironment and the "secretome", i.e., cell signaling molecules and methods. In order to accomplish this study, samples from peripheral or bone marrow blood taken during routine investigations performed during follow-up and re-evaluation visits for the patient's disease as per normal clinical practice will be used. Among the investigations that will be performed on the blood sample will be the genetic/molecular and/or omics and preclinical investigations described above.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be enrolled in the study must have a diagnosis of AML, B ALL/LBL, T ALL/LBL, MPAL/AUL as described by WHO 2016 classification and must complained relapsed or refractory disease after at least one line of therapy
* Ages Eligible for Study: over 18years
* Patients must have greater than 5% blasts in the bone marrow with or without extramedullary disease
* Patients with must have recurrent disease, documented by clinical or radiographic criteria, as well as histologic verification of the malignancy at original diagnosis
* Patients may be enrolled on study regardless of the timing of prior I therapy
* Patients must be capable of understanding the investigational nature and the objectives of the study. All patients must sign a written informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Frequencies of alternative therapies identified for AL patients | 12 months
  Number of patients treated with alternative therapies

OTHER OUTCOMES:
Functional and chemogenomic profiling | 24 months
  Dose-response curves for each drug tested, genetic profile for NGS analyses, description of vesicles contents

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - IRST-IRCCS Meldola, Meldola, Forlì-Cesena
  - A.O.U. Bologna, Bologna
  - A.O.U. Ferrara, Ferrara
  - AOU Parma, Parma
  - Piacenza Hospital - AUSL Piacenza, Piacenza
  - Ravenna Hospital - AUSL Romagna, Ravenna
  - A.O. Reggio Emilia, Reggio Emilia
  - Rimini Hospital-AUSL Romagna, Rimini